CLINICAL TRIAL: NCT06707051
Title: Comparison of Efficacy of Tranexamic Acid and Calcium Dobesilate for Bleeding of Endometrial Origin
Brief Title: Effect of Tranexamic Acid and Calcium Dobesilate for Bleeding of Endometrial Origin
Acronym: TXA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: District Headquarters Teaching Hospital Sahiwal (Other)
Responsible Party: Principal Investigator, Mahpara Shaukat, associate professor, District Headquarters Teaching Hospital Sahiwal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2096; DHQTHS (Other: DHQTHS)
Record Dates: First submitted 2024-10-27; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Heavy. Mentrual Bleeding; Abormal utèrine Bleeding; Bleeding; Uterine Bleeding; Hypersensitivity Response; GI Disturbance; Agranulocytosis; Bleeding Pattern; Endometrial; Endometrial Bleeding
Keywords: Tranexamic acid; Calcium Dobesilate; Bleeding of endometrial origin; TXA
MeSH Terms: conditions — Hemorrhage; Uterine Hemorrhage; Agranulocytosis | interventions — Tranexamic Acid; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): Group A included 50 Patients fulfilling the inclusion and exclusion criteria, was given Tranexamic acid for bleeding of endometrial origin
  Interventions: Drug: Tranexamic Acid
- Group B (Experimental): Group B included 50 Patients fulfilling the inclusion and exclusion criteria, was given Calcium Dobesilate for bleeding of endometrial origin
  Interventions: Drug: Calcium dobesilate (Doxium)

INTERVENTIONS:
Drug: Tranexamic Acid — Group A received Trannexamic Acid 500mg three times a day for 5 days
  Arms: Group A
Drug: Calcium dobesilate (Doxium) — Group B recieved Cap.Calcium Dobesilate 500mg 3 times a day for 5 days
  Arms: Group B

SUMMARY:
Abnormal uterine bleeding is characterized by excessive menstrual blood loss affecting over 50% of women of reproductive age. It can be debilitating and significantly affect a woman's quality of life. Tranexamic acid (TXA) prevents the breakdown of clots and fibrinolysis by binding to the lysine receptor on plasminogen while Calcium dobesilate improves microcirculation and vascular health by increasing nitric oxide synthesis leading to endothelium relaxation, so inhibits endothelial shedding. Calcium dobesilate and tranexamic acid have roles in managing bleeding disorders, but their use and efficacy can vary. Tranexamic acid is more established and widely used for abnormal bleeding, while calcium dobesilate role is less defined and more variable. Tranexamic acid reduces menstrual blood loss, but it has no affect on endothelium while calcium dobesilate reduces the oxidative stress , so improving endothelial health and provide the endothelial protection. Side effects include GI upset , hypersensitivity reactions and agranulocytosis. The side effects of both drugs are comparable.

DETAILED DESCRIPTION:
This Randomized control trial was conducted at Obstetrics & Gynaecology unit Sahiwal Teaching Hospital from to for the period of two years after taking the approval from Institutional review board (IRB). Sample size of one hundred patients (Fifty in each group) was calculated. These patients were randomly allocated into two equal groups, fifty patients in each group. Written informed consent was obtained from each subject by explaining the risks and benefits associated with the drugs. Group A women were given 500mg tranexamic acid thrice a day for 5 days during menstrual cycle and in group B women were given 500 mg capsule Calcium dobesilate thrice a day for 5 days during menstruation for consecutive time period of three months. Women were also evaluated for adverse effects. The information was entered into specially designed proformas. The data was analyzed by SPSS version 21.0. Frequencies and percentages of categorical variables including marital status, parity and adverse effects were calculated and compared between two groups by applying chi square tests. t-Test was used for the calculation of mean and standard deviations of numerical variables like age, BMI, duration of symptoms, blood loss before and after intervention and reduction in blood loss and was compared between two groups. In all statistical analysis only p value less than 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Women of 18-40 years
* Abnormal uterine bleeding

Exclusion Criteria:

* Patients with pregnancy
* Miscarriage
* Hypersensitivity to pharmacological agents to be used in trial
* Patients having moderate to severe anemia (Hb:<8gm/dl)
* Patients with thyroid abnormalities (TSH > 5mIU)
* Benign uterine conditions e.g. fibroid uterus, endometrial/cervical polyp
* Uterine malignancy
* Coagulation disorders (PT : >15sec).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction in blood loss | Three months
  Blood loss at baseline and three months after treatment will measured. Reduction in blood loss will be calculated after three months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sahiwal teaching Hospital Sahiwal, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patient privacy

REFERENCES:
- [Result] Alaqzam TS, Stanley AC, Simpson PM, Flood VH, Menon S. Treatment Modalities in Adolescents Who Present with Heavy Menstrual Bleeding. J Pediatr Adolesc Gynecol. 2018 Oct;31(5):451-458. doi: 10.1016/j.jpag.2018.02.130. Epub 2018 Mar 8. PMID 29524595
- [Result] Klebanoff JS, Marfori CQ, Ingraham CF, Wu CZ, Moawad GN. Applications of Tranexamic acid in benign gynecology. Curr Opin Obstet Gynecol. 2019 Aug;31(4):235-239. doi: 10.1097/GCO.0000000000000547. PMID 31022078
- [Result] Franz ND, Machado-Aranda D, Miller JT, Farina N. Impact of Obesity on Tranexamic Acid Efficacy in Adult Patients With Major Bleeding. Ann Pharmacother. 2021 Sep;55(9):1076-1083. doi: 10.1177/1060028020983323. Epub 2020 Dec 31. PMID 33384016
- [Result] Rahman S, Khan FS, Samin KA, Afridi N, Ahmed M. Efficacy of Oral Tranexamic Acid Versus Combined Oral Contraceptives for Heavy Menstrual Bleeding. Cureus. 2021 Oct 29;13(10):e19122. doi: 10.7759/cureus.19122. eCollection 2021 Oct. PMID 34858760